CLINICAL TRIAL: NCT02942719
Title: The Establishment and Application of the New Labor Progress Centered System of Reducing Cesarean Section Rates in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai First Maternity and Infant Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: FMIH Duan
Record Dates: First submitted 2016-10-18; First posted 2016-10-24 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-10

CONDITIONS: Pregnancy Complications; Postpartum Hemorrhage
MeSH Terms: conditions — Pregnancy Complications; Postpartum Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (20):
- Shanghai First Maternity and Infant Hospital
- Dalian Maternity and Child Health Hospital
- Beijing Obstetrics and Gynecology Hospital
- Shijiazhuang Obstetrics and Gynecology Hospital
- The Children and Women's Healthcare of Laiwu City
- Suzhou Municipal Hospital
- Wenling Women's and Children's Hospital
- First Affiliated Hospital of Kunming Medical University
- Changsha Hospital for Maternal and Child Health Care
- Xinxiang Maternity and Child Health Hospital
- Yanshi People's Hospital
- The Maternal and Child Health Hospital of Guangxi
- Northwest Women and Children's Hospital
- Suining Central Hospital
- Inner Mongolia Maternity and Child Health Hospital
- Fujian Province Maternity and Child Health Hospital
- Qinghai Red Cross Hospital
- Xinjiang Maternity and Child Health Hospital
- Jiangmen Maternity and Child Health Care Hospital
- Gansu Provincial Maternity and Child-care Hospital

SUMMARY:
1. To describe the average labor curve and establish new labor progression standards.
2. Cesarean section rates: Based on big data, the investigator will introduce the international advanced Robson class method and identify the appropriate level of cesarean section rate for each type population.
3. Establishment of "Chinese maternal-fetal medical collaboration network" and APP to promote natural childbirth.

DETAILED DESCRIPTION:
1. To describe the average labor curve and establish new labor progression standards. The investigator will investigate the current characteristics of obstetric population and the labor progression with obstetric intervention in China. The investigator compare the different effects of traditional labor progression management model, new labor progression management model and active labor progression management model on labor outcomes. Based on the best outcomes of maternity and infants, the investigator will establish and modify new labor progression which is suitable for Chinese.
2. Cesarean section rates: Based on big data, the investigator will introduce the international advanced Robson class method and identify the appropriate level of cesarean section rate for each type population.the investigator compare cesarean section rates of different level hospitals and evaluate the effects of reducing cesarean section rates. The investigator also analyze the risk factors of cesarean section rates of the ten Robson classification, which will provide basis for reducing cesarean section rates under the new strategy.
3. Establishment of "Chinese maternal-fetal medical collaboration network" and mobile application software (APP) to promote natural childbirth: The investigator establish perinatal data center using the hospital information system (HIS) system of hospital. The investigator predict the cesarean section rates and relative factors using the Robson classification method, and propose the new strategy of reducing cesarean section rates. Meanwhile, the investigator develop the quality management system toolkit which can help clinicians standardize behavior and improve obstetric safety.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese pregnant women
2. singleton
3. head position
4. 37 weeks + 0 day - 41weeks + 6 days
5. primipara
6. low-risk pregnancy
7. vaginal delivery willingness
8. vaginal cervix <7 cm after labor

Exclusion Criteria:

1. multiple pregnancy
2. non-head position
3. stillbirth
4. selective cesarean section
5. prenatal cesarean section
6. age <18 years
7. previous childbirth history
8. pregnancy complications
9. important fetal malformations.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 20 hospitals from different places of China participated this study. Their annual delivery amount are more than 5000 times and their cesarean section rates are about 40%. The labor progression study include a total of 15,000 puerperae.
Sampling Method: Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
times of uterus contraction | 10 minutes
  The investigator count the times of uterus contraction in 10 minutes both intrapartum and postpartum.

SECONDARY OUTCOMES:
fetal heart rate | 1 minute
  Normal resting fetal heart rate is approximately 120-160 times per minute.
blood pressure | 10 minutes
  Blood pressure is the pressure exerted by circulating blood upon the walls of blood vessels. It is usually expressed in terms of the systolic (maximum) pressure over diastolic (minimum) pressure and is measured in millimeters of mercury (mmHg). Normal resting systolic (diastolic) blood pressure in an adult is approximately 120 mmHg (80 mmHg), abbreviated "120/80 mmHg".
Apgar scores | 1 minute and 5minutes
  The Apgar scale is determined by evaluating the newborn baby on five simple criteria on a scale from zero to two, then summing up the five values thus obtained. The resulting Apgar score ranges from zero to 10.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Duan, Ph.D, Principal Investigator — Shanghai First Maternal and Infant Health Hospital affiliated to Tongji University Medical School
Locations (1):
- Shanghai First Maternity and Infant Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
There are 20 hospitals participated this study, we need get their agreement to share data.